CLINICAL TRIAL: NCT07293689
Title: PREcision MEDicine In Achalasia - A Multicenter Randomized Non-Inferiority Clinical Trial of Short Tailored POEM vs. Standard POEM for Non-Spastic Achalasia and A Multicenter Prospective Cohort Study of Long Tailored POEM for Spastic Esophageal Motility Disorders
Brief Title: PREcision MEDicine In Achalasia (PREMEDIA) - Cohort
Acronym: PREMEDIA
Status: Not yet recruiting | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, John Pandolfino, PRINCIPAL INVESTIGATOR (Contact PI), Northwestern University
Other Study IDs: PREMEDIA (Pro00083748) - 02
Record Dates: First submitted 2025-12-17; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Type III Achalasia; EGJ Outflow Obstruction With Spastic/Hypercontractile Features; Jackhammer Esophagus; Distal Esophageal Spasm
Keywords: achalasia; EGJOO
MeSH Terms: conditions — Esophageal Achalasia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to learn about how the doctor decides how long to cut t the esophageal muscle during Per-Oral Endoscopic Myotomy (POEM) in patients with difficulty swallowing due to certain conditions. The main question it aims to answer is: does pre-POEM testing help the physician choose how long to cut the muscle.

Participants will allow researchers to access their standard of care information in their medical record, complete questionnaires at up to 6 times over a 2-year period.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18
2. Type III achalasia or EGJOO with spastic/hypercontractile features or Jackhammer Esophagus or Distal Esophageal Spasm
3. Eckardt Score > 3

Exclusion Criteria:

* Exclusion:

  1. Prior POEM
  2. Prior surgical treatment for achalasia
  3. Endoscopic pneumatic dilation or lower esophageal sphincter botulinum toxin (botox) injection within 6 months
  4. Prior unrelated esophageal or upper gastric surgery, including Roux-en-Y gastric bypass and sleeve gastrectomy
  5. Prior endoscopic gastroesophageal intervention for obesity or GERD, such endoscopic sleeve gastroplasty or transoral incisionless fundoplication
  6. Known secondary achalasia related to malignancy (pseudoachalasia)
  7. Known eosinophilic esophagitis
  8. Diverticulum (> 2 cm) in distal esophagus
  9. Megaesophagus
  10. Fibroinflammatory stricture of the esophagus due to any etiology (e.g., peptic, radiation, eosinophilic)
  11. Pregnancy
  12. Standard contraindications to general anesthesia
  13. Standard contraindications to endoscopic myotomy in the esophagus (e.g. untreated varices)
  14. Unwillingness or inability to consent for the study
  15. Anticipated inability to follow protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Achalasia, EGJOO, and other spastic motility disorders are relatively rare and have substantial quality of life implications (see Protocol and Research Strategy for details). Given the prevalence and severity of these conditions, it is uncommon for patients with symptoms to not seek some form of treatment. Thus, we expect much of the recruitment to occur directly from site clinics, which include prominent esophageal motility experts and have robust referral networks, as patients seek care. A review of POEM procedure logs from participating CCs reveals that likely eligible patients are on average about 55-65 years old. We anticipate that the ethnic and racial distribution of our study group will be similar to prior achalasia studies with 25% African American, 10% Hispanic and 65% Caucasian.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2029-05-01 (Estimated); Study Completion 2030-03-01 (Estimated)

PRIMARY OUTCOMES:
Clinical Response-Overall | From enrollment to Year 2
  Clinical Response is defined by the Eckardt score (a 4-item self-report scale measuring weight loss, chest pain, regurgitation, and dysphagia) with no need for retreatment in 2 years.
Clinical Response-by Sex | From enrollment to Year 2
  Clinical Response is defined by the Eckardt score (a 4-item self-report scale measuring weight loss, chest pain, regurgitation, and dysphagia) with no need for retreatment in 2 years.
Clinical Response-by Race | From Enrollment to Year 2
  Clinical Response is defined by the Eckardt score (a 4-item self-report scale measuring weight loss, chest pain, regurgitation, and dysphagia) with no need for retreatment in 2 years.
Clinical Response-by Ethnicity | From Enrollment to Year 2
  Clinical Response is defined by the Eckardt score (a 4-item self-report scale measuring weight loss, chest pain, regurgitation, and dysphagia) with no need for retreatment in 2 years.

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - University of California San Diego, La Jolla, California
  - University of Colorado Denver, Denver, Colorado
  - University of Florida, Gainesville, Florida
  - Adventist Health System/Sunbelt, Inc, Orlando, Florida
  - Emory University, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - Washington University, St Louis, Missouri
  - Weill Cornell Medical College, New York, New York
  - Case Western Reserve University, Cleveland, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor Scott & White Health, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR